CLINICAL TRIAL: NCT02647138
Title: The Effect of White Noise In High Noise Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: MARPAC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1502015935
Record Dates: First submitted 2015-12-08; First posted 2016-01-06 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- White Noise (Experimental): Subject will have white noise machine placed in room.
  Interventions: Other: white noise

INTERVENTIONS:
Other: white noise — exposure to white noise

SUMMARY:
Many patients complain to clinicians that they have difficulty sleeping appears to be due to environmental noise. There is a common perception that acute noises are more troublesome than continuous noises in the effect on individual sleep quality. Therefore the goal is to use a Marpac white noise maker with a continuous noise to see its effect on individuals that have difficulty sleeping in a high noise environment.

DETAILED DESCRIPTION:
Insomnia patients will be recruited based on their perception of high noise in their apartment. The investigators will screen patients during the first meeting using The Mini International Neuropsychiatric Interview 6.0 (MINI 6.0). At baseline, an Insomnia Severity Index will be administered.

The study will consist of a one week baseline period in which noise levels will be monitored using spectral analysis and decibel levels and sleep duration will be recorded using a subjective sleep log and wrist actigraphy for objective measurement. At the end of the first week an Insomnia Severity Index will be administered.

During the second week, a treatment period with a white noise machine using a fixed decibel level will be installed in the bedrooms of the subjects. The room noise will continue to be monitored via spectral analysis as well as decibel levels while the patients are wearing actigraphs and keeping a sleep log. At the end of the second week an Insomnia Severity Index will be administered.

During the third week, the white noise machine will be removed and the rooms will still be monitored for sound via spectral analysis and decibel levels and the subject will wear an actigraph and keep a sleep log. At the end of the third week an Insomnia Severity Index will be administered.

The investigators will use Analysis of Covariance (ANCOVA) with baseline vs. white noise to analyze differences. The investigators will use an Acute Noise Index, in which noise spikes of 2 standard deviations from the mean of the entire nights decibel levels count as a noise event.

Noise levels in subjects bedroom will be collected throughout the study along with subjects sleep activity using an actigraph and sleep log.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for each participant are as follows: Must be between 18 and 100 years old
* No significant psychiatric conditions based on the The Mini International Neuropsychiatric Interview 6.0 (MINI 6.0)
* Not currently using narcotics, psychotropic or hypnotic medications and willing to refrain from using these medications during the course of the study
* Limits caffeine consumption to less than or equal to 2 coffee servings, or equivalent per day before 12 noon
* Limits alcohol intake to 7-drinks per week and less than or equal to 1 drinks on any one night
* Must adjust alcohol consumption to 7-drinks per week and less than or equal to 1 drink on any one night for at least two weeks before study begins, and must not consume alcohol later than 8pm
* Naps less than or equal to 1-hour per week according to subjective report
* For at least 3 times a week a minimum of 30 minute sleep latency or 30 minutes of total nighttime awakening due to subjective elevated noise.

Exclusion Criteria:

* Exclusion criteria for each participant are as follows: Younger than 18 years old or older than 100 years old
* Significant psychiatric conditions based on the The Mini International Neuropsychiatric Interview 6.0 (MINI 6.0)
* Currently using narcotics, psychotropic or hypnotic medications and not willing to refrain from using these medications during the course of the study
* Does not limit caffeine consumption to less than or equal to 2 coffee servings, or equivalent per day
* Does not limit alcohol intake to 7-drinks per week and less than or equal to 1 drinks on any one night , consumes alcohol later than 8pm
* Naps more than 1-hour per week according to subjective report
* Not at least 3 times a week at least 30 minute sleep latency or not 30 minutes of total nighttime awakening due to subjective elevated noise

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Sleep Latency data using the actigraph | Three weeks
  Subjects will have three weeks of sleep latency data using the actigraph and this data will be analyzed and presented.

SECONDARY OUTCOMES:
Sleep Latency data using sleep diaries | Three Weeks
  Subjects will have three weeks of sleep latency data using sleep diaries and this data will be analyzed and presented.
Insomnia Severity Index | Three Weeks
  Subjects will complete an Insomnia Severity Index at the end of each of the three weeks of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ana C Krieger, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College Center for Sleep, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.